CLINICAL TRIAL: NCT03940976
Title: Phase 2 Study of Afatinib in Previously Treated Recurrent or Metastasic Esophageal Squamous Cell Carcinoma With EGFR Overexpression or EGFR Amplification (ESCC-A01)
Brief Title: Afatinib in Previously Treated ESCC With EGFR Overexpression or EGFR Amplification (ESCC-A01)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Clinical Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-A01
Record Dates: First submitted 2019-04-28; First posted 2019-05-07 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: afatinib; EGFR Overexpression; EGFR Amplification
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Afatinib (Experimental)
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Afatinib is orally administered at 40mg Qd of each 28 day cycle.

SUMMARY:
This is a phase 2 trial investigating the effect and safety of afatinib in previously treated recurrent or metastasic esophageal squamous cell carcinoma with EGFR overexpression or EGFR amplification.

ELIGIBILITY:
Inclusion Criteria:

1. Having signed informed consent.
2. Age 18 to 70 years old.
3. Histologically confirmed esophageal squamous carcinoma
4. Immunohistochemistry confirmed EGFR(3+) or EGFR-FISH-amplification or next generation sequencing confirmed EGFR-amplification.
5. Computed tomography (CT) or magnetic resonance imaging (MRI) confirmed unresectable metastasic or recurrent ESCC.
6. Refractory or intolerant to at least one regimen.
7. Measurable disease according to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 21 days before enrollment)
8. Life expectancy of ≥3 month
9. Eastern Cooperative Oncology Group (ECOG) 0-2
10. WBC>3,000/mm3, absolute neutrophil count ≥1500/mm3, platelet>100,000/mm3, Hb>9g/dl，Bilirubin level < 1.5 times ULN，Serum creatinine <1.5 times ULN，ALT and AST<2.5 times ULN ，AKP < 2.5 times ULN ，(≤5 times ULN in patients with liver metastases)(within 7 days before enrollment)
11. No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever>38℃.
12. Good compliance

Exclusion Criteria:

1. Contraindications of afatinib.
2. Unable to take afatinib orally because of esophageal stenosis.
3. Currently receiving other effective regimens.
4. Previous anticipate other clinical trial within 4 weeks before entering this study.
5. No measurable lesions, eg. pleural fluid and ascites.
6. With other malignancy within 5 year, except non-melanoma skin cancer and cervical carcinoma in situ.
7. Heart failure or other sever organ dysfunction, eg. coronary artery disease, myocardial infarction within the last 6 months.
8. Mentally abnormal or disable cognition,including central nervous system (CNS) metastasis.
9. HIV infection, active hepatitis B or hepatitis C.
10. Unstable systemic diseases such as poorly controlled diabetes.
11. Interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or evidence of interstitial lung disease showed in X-ray/CT.
12. Keratitis, ulcerative keratitis or severe dry eye syndrome. Known hypersensitivity to study drug.
13. Pregnancy or lactation period.
14. Active severe infection within 14 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-28 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | Until 30 days after the last treatment
  Number of adverse events of afatinib in patients with ESCC.
Disease control rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Percentage of patients who achieve partial response (PR) or complete response (CR) or stable disease (SD) based on Response Evaluation Criteria In Solid Tumors (RECIST).
Progression free survival | Up to 2 years
  Measure of time from study treatment to disease progression or death
Overall survival | Up to 2 years
  Measure of time from study treatment to patient's death or lost to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Professor, Principal Investigator — Peking University Cancer Hospital and Institute
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Liu C, Chen H, Jiao X, Wang Y, Cao Y, Li J, Zhang X, Sun Y, Zhuo N, Dong F, Gao M, Wang F, Dong L, Gong J, Sun T, Zhu W, Zhang H, Shen L, Lu Z. Clinical efficacy and identification of factors confer resistance to afatinib (tyrosine kinase inhibitor) in EGFR-overexpressing esophageal squamous cell carcinoma. Signal Transduct Target Ther. 2024 Jun 28;9(1):153. doi: 10.1038/s41392-024-01875-4. PMID 38937446